CLINICAL TRIAL: NCT06618404
Title: Establishing the Mental Health Needs of People With Spinal Cord Injury
Brief Title: UK Prevalence of Mental Health After SCI
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Collaborators: Spinal Injuries Association (Unknown); University of Buckingham (Unknown)
Responsible Party: Principal Investigator, Katherine Finlay, Dr Katherine Finlay, Lecturer in Psychology, University of Reading
Other Study IDs: MHSCI
Record Dates: First submitted 2021-08-17; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injuries; Anxiety Disorders; Depression; PTSD; Pain
Keywords: Resilience; Mental health; Adjustment; Chronic pain
MeSH Terms: conditions — Spinal Cord Injuries; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Pain; Psychological Well-Being; Chronic Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention - cross-sectional cohort analysis — Observational

SUMMARY:
Mental health decline after Spinal Cord Injury (SCI) is commonly reported but minimally investigated in the United Kingdom. The current study aims to explore the prevalence and impact of mental health challenges after SCI to establish population norms in the UK. Additionally the current study will aim to identify barriers to and facilitators of mental health support seeking in people with SCI.

DETAILED DESCRIPTION:
A four-phase mixed methods research study will be undertaken. Phase One will be a cross-sectional online survey designed to determine the prevalence of mental health conditions in adults with SCI in the UK assessing resilience, anxiety, depression, pain, life satisfaction, PTSD and coping self-efficacy.

Phase Two will consist of in-depth semi-structured online interviews conducted with approximately twenty people with Spinal Cord Injury who, in the first study, indicated either that the participants had accessed, or had wanted to access mental health services. The two-part interview schedule will be undertaken, covering: 1) core themes surrounding the causes of, changes in, and management of mental health after SCI; and 2) questions relating to participant hopes for and experiences of satisfaction with, access to and efficacy of mental health services, in the context of the mental health service providers which participants currently use or have attempted to access.

Phase Three will consist of in-depth semi-structured online interviews held with approximately twenty 'significant others' (partner/family/friend) of people with Spinal Cord Injury whose family member/partner/friend experience mental health problems. The interview schedule will cover two core themes surrounding: 1) perceptions of the causes and impact of mental health difficulties after SCI on 'significant others'; 2) their experiences of current mental health services provided for participants' partner/family/friend and perceived recommendations and hopes for better management of mental health in participants' family member/partner.

Phase Four will recruit twenty-five people with high resilience (>30 on the CD-RISC-10) to participate in an in-depth semi-structured online interview. This will review participants' thoughts and perceptions about resilience and how it is possible to maintain a high level of resilience whilst living with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria: Phases 1 and 2 (survey and SCI interviews)

* Adults with spinal cord injury
* Adults with cauda equina syndrome

Exclusion Criteria:

* Difficulty with written or verbal English Language comprehension

Inclusion Criteria: Phase 3

- Partner, Spouse, Family member or carer of a person with Spinal Cord Injury

Exclusion criteria:

- Difficulty with verbal English Language comprehension

Inclusion Criteria: Phase 4

- Adults with Spinal Cord Injury who screen as having resilience higher than 30 on the Connor-Davidson Resilience Scale (CDRS-10).

Exclusion Criteria: Phase 4

* Adults with Spinal Cord Injury with resilience lower than 30
* Adults with Spinal Cord Injury who choose not to complete the CDRS-10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with spinal cord injury (Phases 1, 2 and 4) or their 'significant others' (Phase 3)
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | Baseline
  Generalised Anxiety Disorder Scale (GAD-7); minimum score = 0; maximum score = 21; Scores higher than 15 represent severe clinical levels of anxiety.
Depression | Baseline
  Patient Health Questionnaire-9 (PHQ-9); minimum score = 0; maximum = 27; scores over 20 represent severe clinical depression.
Post-traumatic Stress Disorder | Baseline
  Impact of Event Scale-Revised (IES-R); 22 item measure of PTSD; minimum score = 0; maximum score = 88; scores over 33 indicate the clinical cut-off for probable PTSD.

SECONDARY OUTCOMES:
Pain Interference | Baseline
  Multi-dimensional Pain Inventory: Spinal Cord Injury (MPI-SCI) Life Interference Subscale; Minimum interference score = 0; maximum interference score = 120; high scores indicate more problematic interference of pain with life.
Coping Self-efficacy | Baseline
  Coping Self-efficacy scale (CSES); minimum score = 0; maximum score = 50 (the mean for each of the five subscales is then summed).
Resilience | Baseline
  Connor-Davison Resilience Scale-10 (CD-RISC-10); minimum score = 0; maximum score = 100; higher scores indicate greater resilience.
Life Satisfaction | Baseline
  Satisfaction with Life Scale (SWLS); minimum score = 5; maximum score = 35, with higher scores indicating greater satisfaction with life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data from the survey will be shared using https://odc-sci.org
Supporting Information: Study Protocol, SAP
Time Frame: From January 2022, indefinitely
Access Criteria: ODC-SCI membership
URL: https://odc-sci.org

DOCUMENTS (1):
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT06618404/ICF_000.pdf